CLINICAL TRIAL: NCT06214897
Title: An Individually Randomized, Partially Blinded, Controlled Trial of Choline-containing Ready-to-use Supplementary Food (C-RUSF) for Children With Moderate Acute Malnutrition to Reduce Deterioration to Severe Acute Malnutrition Compared to Standard RUSF.
Brief Title: Choline to Prevent SAM in Children With MAM
Acronym: CHOP-MAM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Project Peanut Butter (Other); Kamuzu University of Health Sciences (Other); Balchem Corp (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202308159
Record Dates: First submitted 2023-12-31; First posted 2024-01-22 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Moderate Acute Malnutrition

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The intervention and control sachets of RUSF will be packaged such that investigators, outcomes assessors, and participants/caregivers will not know their identity.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- C-RUSF (Ready-to-use Supplemental Food with added choline) (Experimental): A daily dose of 500 Kcal of RUSF containing 500mg choline will be provided
  Interventions: Dietary Supplement: C-RUSF (Ready-to-use Supplemental Food with added Choline)
- S-RUSF (Standard Ready-to-use Supplemental Food without added choline) (Active Comparator): A daily dose of 500 Kcal of RUSF without choline
  Interventions: Dietary Supplement: S-RUSF (Ready-to-use Supplemental Food without added Choline)

INTERVENTIONS:
Dietary Supplement: C-RUSF (Ready-to-use Supplemental Food with added Choline) — Ready-to-use Supplemental Food with added Choline
  Arms: C-RUSF (Ready-to-use Supplemental Food with added choline)
Dietary Supplement: S-RUSF (Ready-to-use Supplemental Food without added Choline) — Standard Ready-to-use Supplemental Food
  Arms: S-RUSF (Standard Ready-to-use Supplemental Food without added choline)

SUMMARY:
The goal of this clinical trial is to test choline supplementation in children with moderate acute malnutrition in Malawi. The main question it aims to answer is:

Will provision of RUSF with added choline (500mg/day) throughout treatment of moderate acute malnutrition (up to 12 weeks) reduce deterioration to severe acute malnutrition among 6-59 month old Malawian children compared with standard RUSF?

DETAILED DESCRIPTION:
Moderate acute malnutrition (MAM) is common among children worldwide, with a prevalence of 50M and an annual incidence likely 3-5x this number. It is defined by mid-upper arm circumference (MUAC) ≥ 11.5 cm and < 12.5 cm or weight-for-length (WLZ) z-score ≥ -3 and < -2. MAM increases a child's risk of deterioration to severe acute malnutrition (SAM), stunting, death, infectious illnesses, and impaired cognitive development. In Malawi, in the year following MAM treatment, nearly one-third of children will face a repeat episode of MAM, 7-10% will develop SAM, and 4% will die. There is much progress yet to be made toward improving rates of recovery and preventing the worst outcomes for the millions of children suffering from MAM each year.

One potential avenue for improving outcomes in MAM is modification of supplementary foods used for its treatment. Choline is an essential nutrient for human health and development, evidence for which is largely drawn from animal models of choline deficiency in which various somatic and cognitive developmental abnormalities are found. Of the trials that have evaluated choline supplementation in humans, many have focused on the role of choline in brain development and, specifically, how it may help foster improved cognitive development in the setting of various insults, such as fetal alcohol syndrome.

There is also a growing body of evidence describing the many roles choline plays outside of the brain, including in the etiology of malnutrition. Recently, choline deficiency has been implicated in the development of kwashiorkor, an enigmatic form of severe acute malnutrition characterized by pitting edema, dermatitis, hair color changes, and fatty liver disease with inflammation. Animal models of choline deficiency display a remarkably similar phenotype to kwashiorkor. When choline has been given to mice, rats, and dogs with kwashiorkor-like malnutrition, the hallmark features of the disease have resolved. This line of evidence suggests a causal role for choline deficiency in kwashiorkor, proposed mechanisms for which include choline's functions in 1-carbon metabolism, sulfur amino acid recycling, and sparing of the essential amino acid methionine. Methionine is the key deficient amino acid in maize-predominant diets, such as are consumed in Malawi. Choline is most abundant in animal-source foods, precisely those which are lacking in the diets of many rural Malawian children. Kwashiorkor accounts for more than one-third of SAM in Malawi in children under 5 years of age and 80% of MAM deterioration to SAM. If the addition of choline to supplementary foods were demonstrated to reduce deterioration to SAM among children with MAM and thereby promote recovery, this would represent an important advance in MAM treatment.

Despite the data supporting choline's essential role in human health and emerging data on its potential therapeutic role in malnutrition, there are no specifications for choline content in food aid products. Common MAM treatment options, such as corn-soy-blend plus and RUSF contain 50-70mg choline, approximately one-third of the 150-200mg recommended for well children 6mo-3y of age. This does not account for the likely increased demand for choline in the setting of malnutrition.

This will be an individually randomized, investigator-blinded, controlled clinical trial. This trial will be conducted at 10 rural sites in southern Malawi where the co-Principal Investigator, Mark Manary, has run malnutrition treatment clinics for over 15 years. The study will include 1500 children (750 per group) 6-59 months of age with uncomplicated MAM, as defined by mid-upper arm circumference (MUAC) ≥ 11.5 cm and < 12.5 cm and/or weight-for-length z-score (WLZ) ≥ -3 and < -2. Exclusion criteria will be presence of nutritional edema, features of complicated MAM, such as mental status changes or breathing issues, as well as participation in a separate feeding program, known allergy to study food ingredient, intention to move away from catchment area within 3 months, developmental delay, or presence of a chronic severe medical condition such as congenital heart disease. Those who wish to take part will undergo randomization, wherein they will remove a single small opaque envelope from a larger opaque envelope and open it, revealing a colored sticker that will correspond to their study group. Caregivers will receive nutrition counselling, complete questionnaires pertaining to demographic, health history/symptoms, and socioeconomic information, and be provided with a two-week supply of their allotted study food for their child. Participants will receive approximately 500 Kcal/day of either C-RUSF or RUSF until they reach a clinical outcome (i.e., graduate, deteriorate to SAM, fail/remain MAM, transfer to hospital, death, default) or for a maximum of 12 weeks. They will be asked to return to clinic fortnightly for re-assessment of anthropometry, illness symptoms, and re-provision of supplementary food until they reach a study outcome. Participants will undergo MDAT testing at time of MAM outcome as well as 5-7 months after MAM outcome to undergo repeat MDAT testing. A randomly chosen subset of participants will undergo blood spot collection at time of MAM outcome.

ELIGIBILITY:
Inclusion Criteria:

* 6-59 months of age
* uncomplicated MAM (mid-upper arm circumference (MUAC) ≥ 11.5 cm and < 12.5 cm and/or weight-for-length z-score (WLZ) ≥ -3 and < -2)
* availability for the duration of the study with no plan to move from the catchment area of a participating clinic

Exclusion Criteria:

* presence of nutritional edema
* features of complicated MAM, such as mental status changes or breathing issues
* participation in another feeding program
* known allergy to study food ingredient
* intention to move away from catchment area within 9 months
* developmental delay
* presence of a chronic severe medical condition (other than TB or HIV) such as congenital heart disease

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1500 (Estimated)
Dates: Start 2024-03-18 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Percentage of pairwise comparisons with wins of Clinical Benefit, which is a composite of time-to-SAM, graduation, and rate of weight change between enrollment and 4-week follow-up. | 2-12 weeks of supplementary feeding
  Clinical benefit is defined as a composite of time-to-SAM, graduation, and rate of weight change. Each participant randomized to C-RUSF is compared to each participant randomized to S-RUSF. For any two participants, a participant will win, i.e. achieve a better clinical outcome, as determined by assessing the following criteria sequentially, stopping when an advantage for either participant is shown:
  Time-to-SAM: developing SAM faster is worse than slower; tied if not possible to determine.
  Graduation: graduating is better than not graduating; tied if not possible to determine.
  Rate of weight change: more positive rate of weight change is better. Rate of weight change is difference in weight (g) between the second follow-up visit and the enrollment visit, divided by enrollment weight (kg), divided by the (d) time elapsed between visits. If the participant lacks data beyond the first follow-up visit, this data will be used instead.

SECONDARY OUTCOMES:
Deterioration to SAM | 2-12 weeks of supplementary feeding
  Children who meet any criteria for SAM during MAM treatment will be considered to have deteriorated to SAM. These are:
  * mid-upper arm circumference (MUAC) < 11.5 cm
  * weight-for-length z-score (WLZ) < -3
  * Presence of bilateral pitting edema
Graduation | 2-12 weeks of supplementary feeding
  Based on the criteria by which the participant was diagnosed with MAM:
  * If a child qualifies for the study based on MUAC < 12.5 cm, the child must obtain MUAC ≥ 12.5 cm.
  * If a child qualifies for the study based on WLZ < -2, the child must obtain WLZ ≥ -2.
  * If a child has MUAC < 12.5 cm and WLZ < -2, either MUAC ≥ 12.5 cm or WLZ ≥ -2 is required for graduation
Rate of weight change | Across first 4 weeks of supplementary feeding
  g/kg/day. Rate of weight gain is calculated as difference in weight in grams between the second follow-up visit (usually 4 weeks after enrollment) and the enrollment visit, divided by enrollment weight (kg), divided by the time between the second follow-up visit and enrollment visit. If the participant lacks data beyond the first follow-up visit, this data will be used instead of the second follow-up visit data. Participants without a follow-up visit will not have data available for rate of weight gain.
Death | From enrollment to end of participant's engagement (at latest, time of 6-month post-outcome MDAT testing)
  Defined by caregiver report
Deterioration to kwashiorkor | 2-12 weeks of supplementary feeding
  Development of nutritional edema (bilateral pedal pitting edema)
Docosahexaenoic acid (DHA) status | 2-12 weeks of supplementary feeding (at time of MAM outcome)
  DHA as % of serum fatty acids
Malawi Developmental Assessment Tool global z-score | 6 months after MAM outcome
  Age-standardized score, -6 to +6, higher scores are better
Malawi Developmental Assessment Tool global z-score | Within 4 weeks of MAM outcome
  Age-standardized score, -6 to +6, higher scores are better
Rate of mid-upper arm circumference (MUAC) change | Across first 4 weeks of supplementary feeding
  mm/week
Rate of length change | 2-12 weeks of supplementary feeding (until MAM outcome)
  mm/week
Deterioration to marasmus | 2-12 weeks of supplementary feeding
  Development of MUAC < 11.5 cm and/or WLZ < -3
Change in MDAT global z-score | From MDAT near time of MAM outcome to 6-month post-MAM-outcome MDAT visit
  Difference in MDAT global z-score between 6-month post-MAM outcome visit and MDAT global z-score measured within 4 weeks of MAM outcome, more positive scores are better
Malawi Developmental Assessment Tool gross motor sub-domain z-score | 6 months after MAM outcome
  Age-standardized score, -6 to +6, higher scores are better
Malawi Developmental Assessment Tool fine motor sub-domain z-score | 6 months after MAM outcome
  Age-standardized score, -6 to +6, higher scores are better
Malawi Developmental Assessment Tool language sub-domain z-score | 6 months after MAM outcome
  Age-standardized score, -6 to +6, higher scores are better
Malawi Developmental Assessment Tool social sub-domain z-score | 6 months after MAM outcome
  Age-standardized score, -6 to +6, higher scores are better
Malawi Developmental Assessment Tool gross motor sub-domain z-score | Within 4 weeks of MAM outcome
  Age-standardized score, -6 to +6, higher scores are better
Malawi Developmental Assessment Tool fine motor sub-domain z-score | Within 4 weeks of MAM outcome
  Age-standardized score, -6 to +6, higher scores are better
Malawi Developmental Assessment Tool language sub-domain z-score | Within 4 weeks of MAM outcome
  Age-standardized score, -6 to +6, higher scores are better
Malawi Developmental Assessment Tool social sub-domain z-score | Within 4 weeks of MAM outcome
  Age-standardized score, -6 to +6, higher scores are better
Diarrhea | 2-12 weeks of supplementary feeding (until MAM outcome)
  Days, reported by caregiver, safety outcome
Proportion of participations requiring hospitalization | 2-12 weeks of supplementary feeding (until MAM outcome)
  Safety outcome

OTHER OUTCOMES:
MDAT global z-score by age | 6-month post-outcome MDAT visit
  Subgroups: enrollment <12 vs. >=12 months of age, -6 to +6, higher scores are better
MDAT global z-score by MAM outcome status | 6-month post-outcome MDAT visit
  Subgroups: Recovered vs. Other, -6 to +6, higher scores are better

CONTACTS AND LOCATIONS:
Overall Officials: Mark J Manary, MD, Principal Investigator — Washington University School of Medicine
Locations (10):
- Malawi (10):
  - Chikonde Health Center, Chikonde
  - Chipolonga Health Center, Chipolonga
  - Makhwira Health Center, Makhwira
  - Mbiza Health Clinic, Mbiza
  - Milonde Health Center, Milonde
  - Mitondo Health Center, Mitondo
  - Muloza Health Clinic, Muloza
  - Namasalima Health Center, Namasalima
  - Naphimba Health Center, Naphimba
  - Nkhate Health Clinic, Nkhate

IPD SHARING:
Plan to Share IPD: Yes
All collected, de-identified individual patient data
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: within 12 months of primary publication